CLINICAL TRIAL: NCT06489496
Title: Prostate Cancer 18F-PSMA-1007 PET/CT Access Trial
Acronym: PAX
Status: Not yet recruiting | Type: Observational
Sponsor: Alberta Health services (Other)
Responsible Party: Principal Investigator, Dr. Denise Chan, Radiologist, Alberta Health services
Other Study IDs: AlbertaHS
Record Dates: First submitted 2024-06-21; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-1007 PSMA PSMA PET/CT — Each patient will receive an IV injection 18F-PSMA-1007 PET/CT.
  PET/CT Imaging will be conducted beginning 90-120 minutes after an injection of 4 MBq/kg (max 400 MBq +/- 15%) 18F-PSMA-1007 in patients.

SUMMARY:
Primary objective:

• To determine if 18F-PSMA-1007 PET/CT imaging is effective at diagnosing prostate cancers and/or metastases compared to conventional imaging [including CT, MRI, 99mTc-MDP Bone Scans as available].

Secondary Objective:

* To determine safety by evaluating for adverse events
* To determine which conventional imaging is being performed when 18F-PSMA-1007 PET/CT imaging is available

DETAILED DESCRIPTION:
Prostate Cancer is the most frequent cancer in men worldwide and accounts for the second leading cause of cancer-related death in men in the United States. Local tumor invasion into neighboring organs such as the seminal vesicle and bladder with distant metastasis to pelvic lymph nodes and bones are frequent. Determining if tumor spread is local or distant influences therapy decisions. Conventional imaging with CT, MRI and bone scans have been used for staging and diagnosis; however, assessment of metastasis particularly lymph node and bone metastasis has remained unsatisfactory. New imaging approaches, which accurately assess disease, are needed to achieve optimal treatment and improve patient outcomes .

In general, PSMA PET imaging appears to have a diagnostic benefit in patients with biochemically recurrent prostate cancer based on elevated serum prostate specific antigen (PSA) levels and negative conventional imaging such as CT and 99mTc-MDP bone scan. It also appears that PSMA PET may perform better over conventional imaging in the initial staging of patients with high-risk prostate cancer. Comparisons between PSMA PET and conventional imaging have been favorable; however, most of these studies have looked at radiopharmaceuticals 18F-DCFPyL or 68Ga-PSMA-11. Studies performed to date have shown that 18F-PSMA-1007 is like other PSMA radiopharmaceuticals in detecting tumor sites. One systematic review demonstrated 18F-PSMA-1007 changed management in 20% of patients at staging. The expectation is that 18F-PSMA-1007 may also eventually replace conventional imaging in the staging and biochemical recurrence work up as other PSMA PET agents. However, larger prospective studies are needed to strengthen its role.

18F-PSMA-1007 PET/CT imaging is changing the management of prostate cancer and may eventually replace conventional imaging in staging and work up for biochemical recurrence. The purpose of this study is to determine if it can replace current conventional imaging (such as CT, MRI, 99mTc-MDP Bone Scans) in clinical practice. The study will also provide patients in Southern Alberta access to this exam that will help with their patient care management.

'• Prospective Phase 3 trial

* Each patient will receive an IV injection 18F-PSMA-1007 PET/CT. Imaging will be conducted beginning 90-120 minutes after an injection of 4 MBq/kg (max 400 MBq +/- 15%) 18F-PSMA-1007 in patients.
* After the 18F-PSMA-1007 PET/CT acquisition is complete, a CT scan will be performed for attenuation correction and localization in the same in line gantry without patient movement between the two scans.
* The results of the 18F-PSMA-1007 PET/CT will be compared to any prior imaging and pathologic results.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Able and willing to follow instructions and comply with the protocol.
3. Provide written informed consent prior to participation in the study.
4. One of the following:

   * a history of radical prostatectomy for treatment of prostate cancer, and a serum prostate specific antigen (PSA) ≥ 0.2 µg/L
   * a history of radiotherapy, cryotherapy, or brachytherapy for treatment of prostate cancer, and a serum PSA progressively rising to ≥ 2 µg/L (minimum two samples) OR a serum PSA doubling-time of < 9 months
   * a history of biopsy-proven prostate cancer and high-risk features for metastatic disease prior to treatment with radical prostatectomy, radiotherapy, cryotherapy, brachytherapy, or other similar therapy. High-risk features include a Gleason score ≥ 8, serum PSA > 20 µg/L, OR minimum clinical T-stage T3a
   * patients who do not meet criteria 1-3 but in whom a 18F-PSMA-1007 PET/CT scan is expected to provide clinical benefit as determined by a Urologist, Radiation Oncologist, Medical Oncologist, or Nuclear Medicine physician (licensed in Alberta)

Exclusion Criteria:

1. Unable to obtain consent
2. Age less than 18 years.
3. Unable to lie flat for 30 minutes to compete PET/CT imaging.
4. Lack of intravenous access

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with history of prostate cancer for staging or clinically suspected recurrent prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of 18F-PSMA-1007 PET/CT imaging to CT/MRI/Bone scans in identifying prostate cancer and/or metastases | 5 year study, approximately 200 patients/ year.
  calculate sensitivity and specificity 18F-PSMA 1007 PET/CT compared to CT, MRI and bone scans using pathology and follow up as gold standard.

SECONDARY OUTCOMES:
To determine safety by evaluating for adverse events | 5 year study, approximately 200 patients/ year.
  evaluate patient reported side effects during and after injection of 18F-PSMA 1007 while in the department

IPD SHARING:
Plan to Share IPD: No